CLINICAL TRIAL: NCT03309462
Title: Analysis of Re-biopsy Specimens in Advanced Non-small Cell Lung Cancer With Acquired Resistance of Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor Targeted Therapy
Brief Title: Analysis of Re-biopsy Specimens in Advanced NSCLC With Acquired Resistance of EGFR-TKI Targeted Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Endoscope Department, Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201701
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Lung Cancer
Keywords: Next generation sequencing; Re-biopsy; Acquired resistance; Tissue sample; Peripheral blood
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re-biopsy tissue sample (Experimental): The gene testing of re-biopsy tissue sample diagnosed with NSCLC will be performed with NGS using Illumina Miseq squencer and Cobas.
  Interventions: Device: Miseq sequencer
- Peripheral blood sample (Experimental): The peripheral blood sample will be extracted with DNA and performed with NGS using Illumina Miseq squencer and ddPCR.
  Interventions: Device: Miseq sequencer

INTERVENTIONS:
Device: Miseq sequencer — The sequencer will be used to detect the gene mutations of the re-biopsy tissue samples and peripheral blood samples obtained from patients.

SUMMARY:
The objective of the study is to reveal the acquired resistance mechanism of the first and second generation Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR-TKI) in tissue and plasma using Next Generation Sequencing (NGS) and the difference of ctDNA in plasma and DNA in biopsy samples is compared and the consistency of two samples was observed. At the same time, the sensitivity, specificity and the consistency of detecting T790M mutation using ddPCR, Cobas and NGS were compared.

DETAILED DESCRIPTION:
With the deepening of the concept of tumor management, it is necessary to monitor the patient's gene during the course of treatment, especially in patients with acquired resistance of the first generation EGFR-TKI. Re-biopsy can effectively provide tissue samples as a "gold standard" for gene detection samples. While, the plasma circulating tumor DNA (ctDNA) detection is an important sample of gene detection and the treatment when tissue samples cannot be assessed. However, due to tumor heterogeneity and ctDNA detection technique sensitivity, plasma ctDNA and tissue samples of the test results are inconsistent. Therefore, the difference between re-biopsy tissue samples and plasma ctDNA samples will provide strong evidence for the application of plasma ctDNA in TKI-resistant patients.

The study was designed as a prospective and single center study. Fifty patients will be enrolled into the study and the clinical data of patients, including smoke history, cancer history, location, pathology, gene mutation status and so on of the first biopsy samples will be collected and recorded in a case report form. For patients recruited in the study, lesions which were assessed as progressive disease(PD) will be obtained by interventional pulmonology technology. And about 20ml peripheral blood will be collected at the same time. The tissue will be divided into two parts, one part was sent to Pathology Department of Shanghai Chest Hospital and will be processed with paraffin-embedded, and for those diagnosed NSCLC, the other part will be extracted with DNA and performed NGS for the qualified DNA sample and using Cobas to detect the T790M mutation. The matched peripheral blood will also be extracted with DNA and performed NGS and ddPCR.

ELIGIBILITY:
Inclusion Criteria:

1. EGFR mutations were confirmed by molecular pathology.
2. Patients who were treated by the first and the second generation EGFR-TKI.
3. Patients were evaluated PD according to RECIST imaging standard.
4. Patients with functional status score (Performance Status, PS) for 0-2 points according to the Eastern Cooperative Oncology Group (ECOG) .
5. Patients can receive histological / cytological specimens through microsurgical biopsy techniques, including but not limited to transbronchial biopsy (TBB), transbronchial lung biopsy (TBLB), transabonchial needle aspiration (TBNA), CT / ultrasound guided thoracic needle aspiration biopsy (CT / ultrasound guided-TTNA), ultrasound-guided superficial lymph node biopsy.

Exclusion Criteria:

1. Patients received blood transfusion within 1 month.
2. Patients suffering from autoimmune diseases, including but not limited to systemic lupus erythematosus, class of wet arthritis, Sjogren's syndrome.
3. Patients with severe disease is not suitable for medical biopsy.
4. Patients refused to participate in clinical trials.
5. Researchers consider that the patient is not suitable for participating in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Compare the differences of gene mutation between tissue sample and peripheral blood sample by NGS | up to one year
  differences of gene mutation between re-biopsy tissue sample and peripheral blood sample will be tested by NGS

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD, PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Xiong L, Xie F, Zheng X, Li Y, Zhu L, Sun J. Next-generation sequencing of tissue and circulating tumor DNA: Resistance mechanisms to EGFR targeted therapy in a cohort of patients with advanced non-small cell lung cancer. Cancer Med. 2021 Jul;10(14):4697-4709. doi: 10.1002/cam4.3948. Epub 2021 Jun 25. PMID 34173341